CLINICAL TRIAL: NCT04898439
Title: The Effect of Greening the School Environment on the Health of Children
Brief Title: GReen And Healthy Schools
Acronym: GRAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Michelle Plusquin, Assistent professor, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Green_School
Record Dates: First submitted 2021-05-10; First posted 2021-05-24 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Function 1, Social; Cognitive Change; Emotions; Weight, Body; Pollution; Exposure
Keywords: greening of schools; biodiversity; cognition; BMI
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: We have 2 groups: an intervention group that includes children from school that will have more nature in its environment and a control school
Masking Description: Children will know whether their school is having more nature
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green school (Experimental): The children from schools that are being greened will be investigated and compared to the control school. We will measure cognitive function, BMI, black carbon levels and emotional wellbeing.
  Interventions: Other: greening of the school environment
- control school (No Intervention): The children from schools that are not being greened will be investigated and used as a control group. We will measure cognitive function, BMI, black carbon levels and emotional wellbeing

INTERVENTIONS:
Other: greening of the school environment — The school will be greened and biodiversity will be increased. This will be done on the playground and area around the school. Special needs corners for playing, relaxing or gardening will be installed.
  Arms: Green school

SUMMARY:
This project aims to investigate the health effects of making schools greener and more biodiverse. We will mainly focus on cognitive effects, well-being, and BMI. The research hypothesis is that greening schools positively influences the health of children through more exercise and cleaner air.

DETAILED DESCRIPTION:
Spending time in nature has been associated with improved physical and mental health and well-being. Developing nature-based health-promoting interventions such as providing more nature in schools to improve children's well-being will lead to benefits for society in our rapidly urbanizing world. Although the benefits of exposure to nature have been demonstrated, knowledge of integrating exposure to nature into public health guidelines is scarce. The latter requires an interdisciplinary approach that integrates the impact of nature-based interventions both on health and on the cost-effectiveness of interventions. Little is known about the health effect of greening and, in particular, increasing biodiversity in schools and we want to investigate further with this study.

This project, therefore, aims to investigate the health effects of greening primary schools and increasing biodiversity and will mainly focus on the effects on cognition, well-being, and BMI. For this, all children from 4th to 6th grade in the participating schools will be invited to participate in this study (Belgium). This study comprises control schools and intervention schools, the schools are examined before the greening and after the greening.

When the informed consent form is signed by the parents, they complete a questionnaire that assesses the child's diet, physical activity, and general questions. A urine sample will be taken for the determination of black carbon particles. The child will also perform computer tests measuring different aspects of "cognition". During these tests, we will also look at the eye movements that play an important role in the cognitive ability of the child. To get an idea of a possible effect on BMI, height and weight will be measured. The child fills in a welfare questionnaire and a questionnaire about the perception of nature itself.

ELIGIBILITY:
Inclusion Criteria:

* Being in 4th, 5th, or 6th grade
* Signed informed consent form by a legal representative

Exclusion Criteria:

* No knowledge of dutch

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function | At the baseline, after 6 months and through study completion, an average of 1 year
  We measure the cognitive function of children by means of a battery of tests including: stroop test, Continuous Performance, digit span, digit signal and digit selection. We combine the computer tests with eye tracking to provide information about saccadic gain during the tests. The computer tests provide data on how much time per reaction (msec) was needed or how many digits could be remembered.
Change in wellbeing | at the baseline, after 6 months and through study completion, an average of 1 year
  We measure the emotional wellbeing by means of the Kids screen test that builds a score of 27 points.
Change in anthropometry | at the baseline, after 6 months and through study completion, an average of 1 year
  We measure BMI and waist/hip circumference. They are expressed as kg/m2 and cm.
Change in black carbon levels | at the baseline, after 6 months and through study completion, an average of 1 year
  We measure urinary black carbon levels. They are expressed as particles per mm2.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Plusquin, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
the protocol and pseudonymised data will be shared
Supporting Information: Study Protocol
Time Frame: 1/9/2021 - 30/12/2022
Access Criteria: UHasselt shared drive